CLINICAL TRIAL: NCT06274749
Title: The Effects of Urolithin A Supplementation on Glucose Metabolism in Healthy Adults >= 55 Years Old. A Randomized Triple-Masked Controlled Clinical Trial
Brief Title: Effects of Urolithin A Supplementation on Glucose Metabolism in Healthy Adults 55 >= Years Old: A Randomized Triple-Masked Controlled Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 10001930; 001930-AG
Record Dates: First submitted 2024-02-22; First posted 2024-02-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-09-29

CONDITIONS: Healthy Volunteer
Keywords: Urolithin A; GLUCOSE METABOLISM; Insulin; Muscle Strength; Microbiomes
MeSH Terms: conditions — Insulin Resistance | interventions — 3,8-dihydroxy-6H-dibenzo(b,d)pyran-6-one

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 50% of participants
  Interventions: Dietary Supplement: Placebo
- Urolithin A (Active Comparator): 50% of participants
  Interventions: Dietary Supplement: Urolithin A

INTERVENTIONS:
Dietary Supplement: Urolithin A — Urolithin A (UA) is a widely available dietary supplement devoid of any known sided effects that is reported to improve mitochondrial function. The UA substance used in this investigation is regulated under Generally Recognized as Safe (GRAS) by the US FDA (GRN No. 000791) (https://www.fda.gov/media/120300/download) and is being advertised and sold as an oral supplement. The daily dose (1 gram) and duration (8 weeks) have already been tested in previous clinical trials.
  Arms: Urolithin A
Dietary Supplement: Placebo — The placebo will consist of methylcellulose and will appear identical to the active supplement. The placebo will be provided by the manufacturer of Urolithin A.
  Arms: Placebo

SUMMARY:
Background:

As people age, the cells in the pancreas that produce insulin begin to release less of this hormone, and levels of blood glucose (sugar) rise. This can lead to illnesses such as diabetes. Urolithin A (UA) is a natural nutritional supplement that may improve how the body controls blood glucose.

Objective:

To learn if UA improves levels of insulin and other hormones that help control blood glucose.

Eligibility:

People aged 55 years and older with a body mass index of 27 or higher.

Design:

Participants will have 6 clinic visits over 8 weeks.

Participants will be screened. They will have a physical exam with blood and urine tests and a test of their heart function.

UA gelcaps are taken by mouth every morning at home. Half of participants will take UA. The other half will take a placebo. The placebo looks like the study drug but does not contain any medicine. Participants will not know which they are taking.

Participants will have tests during the study including:

Oral glucose tolerance: Participants will drink a sweet liquid. Blood will be drawn at intervals over the next 3 hours.

Continuous glucose monitor: A sensor with a needle that goes just under the skin will be placed on the upper arm. Participants will wear this sensor throughout the study.

Exercise. Participants will walk on a treadmill while their heart rate, hearth rhythm, and blood pressure are monitored. They will walk in a hallway at normal and fast paces.

Imaging scans of the thigh; scans of the brain are optional....

DETAILED DESCRIPTION:
Study Description:

We hypothesize that supplementation with the nutritional supplement urolithin A (UA) in healthy adults >= 55 years old will; (i) increase insulin secretion by boosting beta cell metabolism of glucose, resulting in increased ATP generation as pyruvate enters the TCA cycle after glycolysis, thereby enhancing early, acute insulin secretion and glucose uptake in skeletal muscle -both of which will lower circulating levels of blood glucose, (ii) boost production and secretion of incretin hormones because their secretion is also dependent on cellular depolarization, (iii) boost mitochondrial function in brain and muscle tissues. (iv) alter gut microbiome. These effects will be examined over an 8-week period. The study will include a Screening Visit and 5 additional study visits.

Objectives:

Primary Objective:

To determine if UA supplementation will increase the rate at which beta cells respond to glucose.

Secondary Objectives:

Investigate if UA alters incretin secretion in response to oral glucose (incretins are secreted only in response to nutrients) and uncover if UA increases brain and skeletal muscle metabolism.

Endpoints:

Primary Endpoint:

To determine if urolithin A supplementation will influence insulin secretion in response to oral glucose at 4 and 8 weeks after supplementation.

Secondary Endpoints:

* To determine if UA supplementation will increase incretin secretion in response to oral glucose at 4 and 8 weeks after the supplementation.
* To determine if UA supplementation will enhance mitochondria respiration, based on p31 spectroscopy by thigh MRI/MRS at baseline and 8 weeks after supplementation.
* To determine if UA will increase brain oxidative metabolism, based on brain MRS at baseline and 8 weeks after supplementation.
* To determine if UA supplementation will alter gut microbiome composition.
* To determine if Uroltihin A supplementation alters the percentage of immune cell types.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availably for the duration of the study.
* Male or female, age >= 55 years.
* Able to speak and read English. (We do not have ready access to interpreters of different languages at the NIA Clinical Unit).
* BMI >= 27.
* Ability to take oral medication and be willing to adhere to the daily regimen.
* Ability to perform walking and treadmill tests without physical limitations.
* In good general health, as evidenced by medical history/physical exam/laboratory results.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* History of diabetes requiring treatment with any glucose lowering drug(s).
* Fasting glucose >= 126 on screening visit.
* Is on treatment with an investigational drug or other intervention within 8 weeks of enrollment.
* Hospitalization within 12 months for myocardial infarction, coronary revascularization or bypass surgery or stroke.
* History of autoimmune disease, e.g., Hashimoto s thyroiditis, Myasthenia Gravis or Rheumatoid Arthritis.
* Uncontrolled thyroid disease.
* Chronic liver disease indicated by medical history or one of the liver enzymes greater than 2 times the normal range.
* History of chronic kidney disease or GFR <60 mL/min/1.73 m^2.
* Anemia (defined as hemoglobin level <12 g/dl for men or < 11 g/dl for women).
* Poor venous access.
* Uncontrolled hypertension as judged by the Investigator.
* History of significant GI disease, e.g., IBS, Crohn s disease.
* Active cancer or has had treatment for cancer in the last 1 year.
* Medical condition requiring absolute and continuous need for long-term treatment with antibiotics, corticosteroids, immunosuppressors.
* Currently pregnant or a nursing mother due to possible changes in hormones and metabolism.
* History of, or laboratory evidence of HIV virus infection at Screening Visit.
* History of, or laboratory evidence of Hepatitis B or C at Screening Visit.
* Positive urine drug screen at Screening Visit (unless taking prescribed medication and at the discretion of the PI).
* Reports claustrophobia and/or is not eligible to have an MRI as per the MRI eligibility form.
* Weight >= 300 lbs (MRI scanner weight limit).
* Hip or knee replacement or other medical condition that prevents MRI research scans from being performed.
* Diagnosed with cognitive impairment that clearly prevents the participant from providing informed consent.
* Current smoker or tobacco use in the past year.
* History of substance abuse, including marijuana use in the past year.
* On average, consumes more than 1 alcoholic drink per day.
* Any other condition which in the investigator s opinion may adversely affect the subject s ability to complete the study or its measures or which may pose significant risk to the subject.

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
To determine if urolithin A supplementation will influence insulin secretion in response to oral glucose at 4 and 8 weeks after supplementation. | 8 weeks
  Study visits 1 - 5

SECONDARY OUTCOMES:
To determine if UA supplementation will increase incretin secretion in response to oral glucose at 4 and 8 weeks after the supplementation. | 8 weeks
  Study visits 1 - 5
To determine if UA supplementation will enhance mitochondria respiration, based on p31 spectroscopy by thigh MRI/MRS at baseline and 8 weeks after supplementation. | 8 weeks
  Study visits 1 & 5
To determine if UA will increase brain oxidative metabolism, based on brain MRS at baseline and 8 weeks after supplementation. | 8 weeks
  Study visits 1 & 5
To determine if UA supplementation will alter gut microbiome composition. | 8 weeks
  Study visits 1, 3 & 5

CONTACTS AND LOCATIONS:
Overall Officials: Josephine M Egan, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001930-AG.html